CLINICAL TRIAL: NCT02585089
Title: Beneficial Effects of Pork Bioactive Peptides on Cardiovascular Health in Humans
Brief Title: Effects of Cured Pork Peptides on Blood Pressure & Cardiovascular Risk Factors
Acronym: PocPep-CVD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, LUIS TEJADA PORTERO, Lecturer, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: UCAM-BACCHUS
Record Dates: First submitted 2015-07-31; First posted 2015-10-23 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Hypertension; Cardiovascular Diseases
Keywords: Hypertension; active biopeptide; cardiovascular pathophysiology; angiotensin converting enzyme inhibition; cured-pork ham
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spanish cured-pork ham (Active Comparator): One group will receive dry-cured pork ham of >10 months proteolysis (intervention product).
  Intervention: Dietary intake Dry-cured pork ham contains high doses of bioactive peptides produced during more than 10 months of proteolysis.
  Interventions: Other: Spanish cured-pork ham
- Cooked pork ham (Placebo Comparator): The other group will receive cooked, uncured ham (placebo product). Intervention: Dietary intake. Cooked ham does not display bioactive peptides as they are produced during proteolysis of pork ham.
  Interventions: Other: Cooked pork ham

INTERVENTIONS:
Other: Spanish cured-pork ham — Dry-cured ham with reduced salt will be used in order to decrease the sodium intake that could affect blood pressure too. Such ham contains 25% lower salt than similar products on the market (3,7g vs 4,5g/100g).
  Volunteers will receive 80g of cured pork ham daily for 28 consecutive days. They can eat the interventional product at any time of the day.
  Arms: Spanish cured-pork ham
Other: Cooked pork ham — Volunteers will receive 100g of cooked pork ham daily for 28 consecutive days. They can eat the product (placebo product) at any time of the day.
  Arms: Cooked pork ham

SUMMARY:
Spanish dry-cured ham has been shown a source of antihypertensive peptides in mice. To date, no clinical study has been performed in humans to check the effects of bioactive peptides produced naturally during the processing of pork dry-cured ham on blood pressure. Therefore, the aim of the present study is to investigate whether consuming peptides from cured pork ham with demonstrated angiotensin I-converting enzyme (ACE) inhibitory activity lowers blood pressure (BP) and improves other risk factors for cardiovascular disease (CVD).

Objectives: To demonstrate the lowering effects of bioactive peptides from cured pork ham with >10 months dry-curing process in humans. To check for other possible benefits related to dry-cured ham intake such as: platelet activation and cardiovascular risk factors.

DETAILED DESCRIPTION:
A two-arm cross-over clinical study with a diet control will be assessed at the Catholic University of Murcia (UCAM).

A recruitment of 50 volunteers will be attempted in order to fulfil the UCC calculations. The 50 patients will be divided into two groups (25 vs 25). One group will receive dry-cured pork ham of >10 months proteolysis (intervention product) while the other will receive cooked, uncured ham (control product), each for one month. After two weeks wash out, the groups will be exchanged for one additional month. In this way, each group will take cooked ham and dry-cured pork ham for 28 days each arm.

Pork hams Two pork hams from the same raw meat will be used in the present study: dry-cured pork ham with >10 months dry-curing process as the intervention product and cooked, uncured ham as the control product. Both products will be purchased in vacuum bags and labelled with safety information (expiration date, nutritional composition and storage information).

Dry-cured ham with reduced salt will be used in order to decrease the sodium intake that could affect BP too. Such ham contains 25% lower salt than similar products on the market (3,7g vs 4,5g/100g) (see leaflet of a possible ham enclosed).

Dry-cured ham (80g) will be taken daily by the volunteers (50% humidity); BP will be measured as follows. In order to counteract the higher water contain (70% humidity), a higher amount of cooked ham will be given to the control groups (100g). Besides, cooked ham contains 2.5g salt/100g which is in relation with the 2,96g salt/80g reduced salt dry-cured ham. A restriction list food will be also given to the volunteers in order to control salt intake.

Volunteers Caucasian men and women, aged 35-60 years, in good general health with an average of systolic arterial pressure >130 mmHg and diastolic > 80 mmHg will be recruited. Exclusion criteria are: smokers, Diabetes mellitus, diagnosed and treated hypertension, history of cardiovascular events (stroke, myocardial infarction or peripheral vascular disease), medications: anti-hypertensives, vasodilators, lipid lowering therapies and fish oil supplements unless willing to discontinue prior to and during study (all other supplements will be assessed on a case by case basis).

Weight, height, body mass index and waist circumference will be measured at the beginning of the study by qualified nurses. A list of restricted food will be given at the beginning of the study in order to avoid excessive salt consumption.

Besides, three 24h intake surveys will be conducted for three no consecutive days (one of them on Sunday) during the study. Another survey regarding their diet habits and salt intake will be also conducted three times, once with each ham and in wash out period.

Blood pressure measurements Blood pressure will be measured with two different approaches: 24h ambulatory monitoring of BP.

24h ambulatory monitoring. A 24h recording will be assessed to all the volunteers included in the study at four different time points (before/after control product and before/after intervention product). Volunteers will be appointed for a blood extraction and a digital manometer device OMRON M24/7 BP5 properly calibrated will be installed to each volunteer.

Home auto-monitoring of BP. Auto-measurement of BP will be performed following the recommendations of the Spanish Society of Hypertension, Spanish League Against Hypertension (SEHLELHA) and the European Society of Hypertension (ESH) three times during each intervention. On the day of first appointment at the doctor office, individuals will be taught how to auto-measure its BP at home and the dominant arm will be determined. A digital manometer device OMROM 705CP properly calibrated will be given to each volunteer for a short period of time. BP will be measured 3 times during each interventional product (cured pork ham and cooked ham) as follows. The three different days, the volunteer will be asked to measure three times per day (before breakfast, 2h after pork consumption -preferably before lunch- and before dinner), and each measurement will be repeated for three times, about one minute apart. The volunteer will measure its BP seated after resting 5 min in this position, he will not smoke, ingest food or caffeine beverages (coffee, tea or colas), or exercise (including stair climbing) in the previous 30 minutes prior to the time of measurement. Measurements will be done in the dominant arm. The systolic and diastolic blood pressure readings will be recorded. The mean of the three measures will be used for all analyses.

Biochemical parameters Blood will be taken before each phase (cured pork ham/cooked ham) and after the end of such intakes, following by a 2 weeks wash out period (total 4 time points). Blood analysis will be performed after fasting for at least 8 hours.

Blood lipid profile (total cholesterol, HDL, LDL and triglycerides); hemogram, plasma glucose, creatinine, albumin and uric acid will be measured.

Plasma will be collected and stored at -80ºC for further analysis such as C reactive protein, fibrinogen and interleukins if the case.

Participants will be asked to provide a 24-hour urine collection and they will be given written and verbal instructions for the 24-hour collection. The first urine of the day will be discarded and all urine over the following 24 hours will be collected in standard containers that will be provided. Total volume of the collection will be measured by the volunteers. Urine collections will be rejected if 24-hour urinary volumes were less than 250 mL, or if the timing of the collection fell outside the range of 20-28 hours. In accordance with the standard procedure, urinary sodium and potassium will be measured using ion selecting electrode method.

Daily salt intake will be estimated based on calculation of 24-hour urinary sodium excretion on the assumption that all sodium ingested was in the form of sodium chloride.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men and women,
* aged 35-60 years in good general health with an average of systolic arterial pressure >130 mmHg and diastolic >80 mmHg.

Exclusion Criteria:

* smokers,
* Diabetes mellitus,
* diagnosed and treated hypertension,
* history of cardiovascular events (stroke, myocardial infarction or peripheral vascular disease),
* receiving medications: anti-hypertensives, vasodilators, lipid lowering therapies and fish oil supplements unless willing to discontinue prior to & during study (all other supplements will be assessed on a case by case basis).

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Systolic Blood Pressure at 28 days | Before/after 28 days of interventional product and placebo product
  24h holters (OMROM) will be used for comparing blood pressure during the study

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Zafrilla, PhD, Study Chair — UCAM
Locations (1):
- Catholic University of Murcia (UCAM), Murcia, Murcia, Spain

REFERENCES:
- See also: Related Info — http://www.bacchus-fp7.eu/